CLINICAL TRIAL: NCT00662012
Title: Sodium Stibogluconate Treatment of Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-10950; WU#01-19002 (Other: WRAIR)
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Leishmaniasis
Keywords: Leishmaniasis; Sodium stibogluconate; Pentostam; sand fly
MeSH Terms: conditions — Leishmaniasis | interventions — Antimony Sodium Gluconate; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Stibogluconate (SSG) 20 mg/kg (Experimental): All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with 20 mg/kg once daily intravenously with SSG.
  Interventions: Drug: Sodium Stibogluconate (SSG)

INTERVENTIONS:
Drug: Sodium Stibogluconate (SSG) — 100 mg/ml/vial. Treatment for laboratory-confirmed leishmaniasis with SSG 20mg/kg/d intravenously (IV) for 10 days or 20 days for less responsive; visceral leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days as a second line of therapy for those failing or intolerant of Ambisome; and mucosal leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days.
  Other Names: Pentostam (GlaxoSmithKline)

SUMMARY:
Leishmanias is a disease caused by the bite of sandflies and is found in many parts of the world including the Europe, Southwest Asia, Africa and the Middle East. This disease is a threat for military soldiers in areas where this disease is found. Sodium stibogluconate (SSG) or Pentostam (Glaxo Smith Kline, United Kingdom) is an Investigational New Drug (IND) product used by the Department of Defense for over 20 years to treat cutaneous, mucosal and viseral leishmanias. This drug is not licensed for commercial use in the United States because of very limited need for the product in the U.S.A. The objective of this protocol is to provide sodium stibogluconate for the treatment of cutaneous leishmaniasis and mucosal leishmaniasis (pentavalent antimonials curently considered the drug of choice for these infections) Provide sodium stibogluconate as a second line treatment for viscerotropic and visceral leishmaniasis (liposomal amphotericin is the drug of choice for these types as it is FDA approved for vusceral leishmaniasis).

DETAILED DESCRIPTION:
Leishmaniasis is a protozoal disease transmitted by sandflies and is endemic in many parts of the world including Central and South America, Europe, Southwest Asia, Africa, and the Middle East. Infected humans may develop cutaneous (Old or New World), mucocutaneous (New World), or visceral leishmaniasis. The disease is a medical threat for military soldiers assigned in endemic areas and currently a major cause of morbidity in soldiers deployed to the Middle East and a complication of military exercises in Panama, Honduras, and South America.

Pentavalent antimonials (Pentostam, GSK, UK, and Glucantime, Rhone-Poulenc, France) have been used to treat leishmaniasis for more that 50 years. Neither of these drugs are licensed for commercial use in the United States, likely because of limited use. Worldwide, there is a great deal of experience and use of these products.

Pentostam or sodium stibogluconate is a pentavalent antimony drug complexed to carbohydrate the exact structure and mechanism of action of which are not known. It is provided as a 100 mg antimony/ml solution that contains a preservative, m-chlorocresol. Most of the dose is excreted by the kidneys within 24 hours.

Pentostam is presently an investigational new drug (IND) product that has been in use by the Department of Defense (DoD) for over 20 years for the treatment of cutaneous, mucosal and visceral leishmaniasis. In August, 1997, the FDA approved Ambisome (liposomal amphotericin) for the treatment of visceral leishmaniasis. As a result, in the treatment of visceral and viscerotropic leishmaniasis, the use of antimonials will now be considered a second-line therapy

In 1984, the World Health Organization recommended that the daily dose of antimony in the treatment of visceral leishmaniasis be increased to 20 mg/kg/day. A randomized controlled trial of 40 subjects with American, New World, cutaneous leishmaniasis (ACL) found 100% cure rates with 20 mg/kg/day Sb for 20 days but only a 76% cure if 10 mg/kg/day for 10 days was used. A comparison of three treatment schedules in 36 subjects with CL (single rapid infusion, continuous 24 hour infusion, or every eight hour doses) found no advantage over using once daily dosing. A review of the controlled trials of SSG concludes that a recommended course of therapy is 20 mg/kg/day with no upper limit to dose for 20 days for CL and 20 mg/kg/day for 28 days for visceral or mucocutaneous leishmaniasis. The Pentostam® package insert suggests that 10-20 mg/kg/day with a maximum dose of 850 mg for a minimum of 20 days be used; however, based on the Centers for Disease Control and Prevention (CDC) and Walter Reed Army Medical Center (WRAMC) experience and their practice guidelines, 20 mg/kg/day with no upper limit to dosage is used. WRAMC recently published their CL treatment experience primarily in New World leishmaniasis comparing SSG 20 mg/kg for 10 or 20 days and found 100% of volunteers in the 10-day group were cured. In this study 15% were Leishmania major infections. Comparable results are expected for Old World leishmaniasis based on clinical experience and current literature.

Detailed toxicity data for the 20 mg/kg/day dose are provided by several studies. Percentages from the WRAMC experience are included here. Subjective musculoskeletal complaints are common (58%), as well as elevated hepatocellular (67%) and pancreatic enzyme levels (97%) and nonspecific electrocardiogram (EKG) changes (T wave changes). These side effects are usually reversible, and no deaths have been associated with SSG at WRAMC. Other SSG toxic effects include headache (22%), rash (9%), thrombocytopenia, depression of various hematologic cell lines (44%), phlebitis, anaphylaxis, inflammation around lesions, and transient coughing after infusion. Other associated symptoms include anorexia, malaise, myalgia, abdominal pain, headache, lethargy, sweating, vertigo, facial flushing, initial worsening of skin lesions, epistaxis, jaundice and peripheral neuropathy. In our above-mentioned 10 versus 20 days study, the adverse events (AE) were significantly decreased in the cohort receiving the 10 days versus 20 with myalgias in 42% (versus 68%), with less chemical pancreatitis and fewer hematologic parameter disorders. Angioedema during SSG infusion has recently been described in two subjects at WRAMC. Both subjects responded quickly to benadryl treatment without complications. Both subjects were subsequently skin tested with SSG intradermally for hypersensitivity and one reacted.

Alternative heat therapies have been used to successfully treat CL. Laboratory investigation showed that Leishmania infection is sensitive to heat. Various forms of heat application in human CL has shown variable efficacy. The TTI Thermomed™ device has been cleared as a 510-k device by the U.S. Food and Drug Administration (FDA) for use in the treatment of CL. This device uses localized current field radio frequency. Other therapies that may be effective for treating CL include topical paromomycin and oral fluconazole.

ELIGIBILITY:
Inclusion Criteria:

* DoD healthcare beneficiary of any age and gender.
* Clinicoepidemiologic or parasitologic diagnosis (microscopy, PCR or culture) of Leishmania infection.
* Able to provide informed consent or assent (children).
* All participants (both male and female) must agree to take precautions not to become pregnant or father a child for at least 2 months after receiving SSG.

Exclusion Criteria:

* Pregnancy. Females of childbearing potential must have negative urine human chorionic gonadotropin hormone (HCG) within 96 hours start of infusion period.
* History of hypersensitivity to pentavalent antimonials.
* Any of the following on screening examination:

  1. QTc interval greater or equal to 0.5 sec
  2. Severe cardiac disease (disabling valvular heart disease, myopathy, or arrhythmias)
  3. History of recurrent pancreatitis
  4. Liver failure or active hepatitis with transaminases > 3x upper limit of normal
  5. Renal failure or creatinine > 2.5 mg/dL
  6. Thrombocytopenia (platelets <100,000/mm3)
  7. White blood cell count < 2000 / mm3
  8. Hematocrit < 30 %

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2002-06; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wortmann, MD, Principal Investigator — Walter Reed Army Medical Center, Infectious Disease
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Walter Reed Army Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment commenced on 11May2002 with follow-up periods ranging from 12 to 24 months after completion of treatment. Treatment was received at Walter Reed Army Medical Center, Washington, DC, USA.
Groups:
- SSG 20 mg/kg: All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with 20 mg/kg once daily intravenously with SSG.
  Sodium Stibogluconate (SSG): 100 mg/ml/vial. Treatment for laboratory-confirmed leishmaniasis with SSG 20mg/kg/d intravenously (IV) for 10 days or 20 days for less responsive; visceral leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days as a second line of therapy for those failing or intolerant of Ambisome; and mucosal leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days.
Period: Overall Study
Arm/Group | SSG 20 mg/kg
Started | 414
Completed | 327
Not Completed | 87
Not completed — Lost to Follow-up | 85
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat, evaluable, and safety populations included all patients who received at least 1 dose of SSG. Data were displayed by regimen and overall for patients with CL.
Arm/Group | SSG 20 mg/kg
Number analyzed (Participants) | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 405
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 62
  White | 295
  More than one race | 0
  Unknown or Not Reported | 50
Region of Enrollment [Number; unit: participants] — All subjects must be willing to locate to the WRAMC area during treatment
  participants
    United States | 414
Lesion data - Duration since onset [Mean (Standard Deviation); unit: Days] | 111.6 (47.62)
Lesion data - Number of lesions [Mean (Standard Deviation); unit: Lesions] — Number of lesions on body
  Lesions | 5.0 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint - Frequency of Complications of Therapy
Description: The primary safety endpoint is the frequency of complications of therapy
Time Frame: 5 years
Population: Analysis was per protocol
Measure: Number; unit: participants
Arm/Group | SSG 20 mg/kg
Number analyzed (Participants) | 414
participants | 414

2. Secondary Outcome: Improvement of Lesions, Resolution of Fever and Lab Abnormalities for Visceral Leishmaniasis and Regression of Mucosal Lesions .
Description: Improvement of lesions for cutaneous leishmanias, resolution of fever and lab abnormalities for visceral leishmaniasis and regression of mucosal lesions for mucocutaneous disease.
Time Frame: 5 years
Population: Analysis per protocol
Measure: Number; unit: participants
Arm/Group | SSG 20 mg/kg
Number analyzed (Participants) | 414
participants | 414

ADVERSE EVENTS:
Time Frame: The study included a screening/baseline period, a 10-20 or 28-day treatment period, and a 12-24 month follow-up period.
Description: 10 days for cutaneous leishmaniasis due to L. major, 20 days for cutaneous leishmaniasis due to other species and for some more severe or less responsive L. major infections, 28 days for mucocutaneious, viscerotripic, or visceral leishmaniasis.
Arm/Group | SSG 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 17/414
Other Adverse Events (participants affected / at risk) | 414/414
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSG 20 mg/kg (N=414)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Meningitis Aseptic (Immune system disorders) | 3 (3)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Calculus Ureteric (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Lymphacele (Vascular disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Gall Bladder Disorder (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cutaneous Leishmaniasis (Infections and infestations) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Heat Exhaustion (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 1 (1)
Road Accident (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Biopsy Liver (Investigations) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Aneurysm Ruptured (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSG 20 mg/kg (N=414)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 21 (21)
Lymphadenopathy (Blood and lymphatic system disorders) | 59 (59)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10)
Bundle Branch Block Left (Cardiac disorders) | 4 (4)
Bundle Branch Block Right (Blood and lymphatic system disorders) | 22 (22)
Conduction Disorder (Cardiac disorders) | 9 (9)
Dilatation Atrial (Cardiac disorders) | 8 (8)
Palpitations (Cardiac disorders) | 9 (9)
Sinus Tachycardia (Cardiac disorders) | 6 (6)
Supraventricular Extrasystoles (Cardiac disorders) | 6 (6)
Tachycardia (Cardiac disorders) | 55 (55)
Ventricular Extrasystoles (Cardiac disorders) | 6 (6)
Ventricular Hypertrophy (Cardiac disorders) | 9 (9)
Ear Pain (Ear and labyrinth disorders) | 4 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 7 (7)
Abdominal Distension (Gastrointestinal disorders) | 15 (15)
Abdominal Pain (Gastrointestinal disorders) | 118 (118)
Abdominal Pain Lower (Gastrointestinal disorders) | 8 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 33 (33)
Abdominal Tenderness (Gastrointestinal disorders) | 20 (20)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 59 (59)
Dyspepsia (Gastrointestinal disorders) | 18 (18)
Flatulence (Gastrointestinal disorders) | 7 (7)
Gastritis (Gastrointestinal disorders) | 7 (7)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 135 (135)
Pancreatitis (Gastrointestinal disorders) | 151 (151)
Stomach Discomfort (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 31 (31)
Asthenia (General disorders) | 4 (4)
Chest Discomfort (General disorders) | 4 (4)
Chest Pain (General disorders) | 21 (21)
Chills (General disorders) | 8 (8)
Early Satiety (General disorders) | 4 (4)
Fatigue (General disorders) | 292 (292)
Feeling Hot (General disorders) | 5 (5)
Infusion Related Reaction (General disorders) | 12 (12)
Infusion Site Reaction (General disorders) | 23 (23)
Oedema Peripheral (General disorders) | 5 (5)
Pain (General disorders) | 9 (9)
Pyrexia (General disorders) | 51 (51)
Thirst (General disorders) | 6 (6)
Hepatitis (Hepatobiliary disorders) | 45 (45)
Cellulitis (Infections and infestations) | 7 (7)
Folliculitis (Infections and infestations) | 7 (7)
Herpes Simplex (Infections and infestations) | 6 (6)
Herpes Zoster (Infections and infestations) | 8 (8)
Pharyngitis (Infections and infestations) | 5 (5)
Rhinitis (Infections and infestations) | 6 (6)
Sinusitis (Infections and infestations) | 7 (7)
Skin Infection (Infections and infestations) | 8 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 74 (74)
Wound Infection (Infections and infestations) | 11 (11)
Alanine Aminotransferase Increased (Investigations) | 245 (245)
Anion Gap Decreased (Investigations) | 6 (6)
Aspartate Aminotransferase Increase (Investigations) | 202 (202)
Blood Albumin Decreased (Investigations) | 53 (53)
Blood Alkaline Phosphatase Increased (Investigations) | 19 (19)
Blood Amylase Increased (Investigations) | 273 (273)
Blood Billirubin Increased (Investigations) | 8 (8)
Blood Calcium Increased (Investigations) | 5 (5)
Blood Chloride Increased (Investigations) | 19 (19)
Blood Glucose Decreased (Investigations) | 25 (25)
Blood Glucose Increased (Investigations) | 29 (29)
Blood Potassium Decreased (Investigations) | 21 (21)
Blood Potassium Increased (Investigations) | 4 (4)
Blood Pressure Increased (Investigations) | 19 (19)
Blood Sodium Increased (Investigations) | 9 (9)
Blood Urea Increased (Investigations) | 7 (7)
Body Temperature Increased (Investigations) | 10 (10)
Electrocardiogram P Wave Abnormal (Investigations) | 6 (6)
Electrocardiogram QRS Complex Abnormal (Investigations) | 12 (12)
Electrocardiogram ST Segment Abnormal (Investigations) | 28 (28)
Electrocardiogram ST Segment Elevation (Investigations) | 11 (11)
Electrocardiogram T Wave Abnormal (Investigations) | 83 (83)
Electrocardiogram T Wave Inversion (Investigations) | 13 (13)
Electrocardiogram Abnormal (Investigations) | 22 (22)
Electrodardiogram Repolarisation Abnormality (Investigations) | 8 (8)
Eosinophil Count Increased (Investigations) | 6 (6)
Eosinophil Percentage Increased (Investigations) | 32 (32)
Haematocrit Decreased (Investigations) | 79 (79)
Haemoglobin Decreased (Investigations) | 21 (21)
Heart Rate Increased (Investigations) | 20 (20)
Lipase Increased (Investigations) | 331 (331)
Lymphocyte Count Decreased (Investigations) | 17 (17)
Lymphocyte Percentage Decreased (Investigations) | 65 (65)
Lymphocyte Percentage Increased (Investigations) | 9 (9)
Monocyte Count Increased (Investigations) | 25 (25)
Monocyte Percentage Increased (Investigations) | 76 (76)
Neutrophil Count Decreased (Investigations) | 11 (11)
Neutrophil Count Increased (Investigations) | 17 (17)
Neutrophil Percentage Decreased (Investigations) | 9 (9)
Neutrophil Percentage Increased (Investigations) | 22 (22)
Pancreatic Enzymes Increased (Investigations) | 6 (6) — The low frequency of event relative to the laboratory data, show a high frequency of increases in pancreatic enzymes,is due to the fact that most abnormalities in pancreatic enzymes were coded to the specific pancreatic enzyme (amylase or lipase)
Platelet Count Decreased (Investigations) | 88 (88)
Protein Total Decreased (Investigations) | 12 (12)
QRS Axis Abnormal (Investigations) | 31 (31)
Red Blood Cell Count Decreased (Investigations) | 16 (16)
Transaminases Increased (Investigations) | 10 (10)
Tuberculin Test Positive (Investigations) | 4 (4)
Urine Antimony Increased (Investigations) | 11 (11)
White Blood Cell Count Decreased (Investigations) | 120 (120)
White Blood Cell Count Increased (Investigations) | 22 (22)
Anorxia (Metabolism and nutrition disorders) | 54 (54)
Decreased Appetite (Metabolism and nutrition disorders) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 286 (286)
Back Pain (Musculoskeletal and connective tissue disorders) | 44 (44)
Flank Pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Groin Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 (8)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 18 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 253 (253)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 5 (5)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Dizziness (Nervous system disorders) | 30 (30)
Dysgeusia (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 212 (212)
Hypoaesthesia (Nervous system disorders) | 6 (6)
Migraine (Nervous system disorders) | 6 (6)
Paraesthesia (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 12 (12)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 42 (42)
Post-traumatic Stress Disorder (Psychiatric disorders) | 4 (4)
Sleep Disorder (Psychiatric disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Dry Skin (Skin and subcutaneous tissue disorders) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7)
Night Sweats (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (17)
Rash (Skin and subcutaneous tissue disorders) | 67 (67)
Rash Papular (Skin and subcutaneous tissue disorders) | 7 (7)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 5 (5)
Skin Lesion (Skin and subcutaneous tissue disorders) | 35 (35)
Urticaria (Skin and subcutaneous tissue disorders) | 10 (10)
Flushing (Vascular disorders) | 7 (7)
Hot Flush (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 23 (23)
Phlebitis (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No